CLINICAL TRIAL: NCT05088967
Title: A Randomized, Open-label, Phase Ib Clinical Study to Evaluate the Efficacy and Safety of IBI110 in Combination With Sintilimab Versus Sintilimab Alone in Neoadjuvant and Adjuvant Therapy of Radically Resectable Non-small Cell Lung Cancer
Brief Title: Efficacy and Safety of IBI110 in Combination With Sintilimab Versus Sintilimab Alone in Neoadjuvant and Adjuvant Therapy of Radically Resectable Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Development strategy adjustment
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI110C201
Record Dates: First submitted 2021-09-28; First posted 2021-10-22 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBI110+sintilimab (Experimental): IBI110 and sintilimab will be administered as intravenous (IV) infusion on Day 1 of each 21-day cycle (every 3 weeks) for 3 cycles during the neoadjuvant treatment phase. IBI110 and sintilimab will be administered as IV infusion 3 weeks during the post-operative adjuvant phase up to 1 year.
  Interventions: Drug: IBI110; Drug: sintilimab
- sintilimab (Active Comparator): Sintilimab will be administered as intravenous (IV) infusion on Day 1 of each 21-day cycle (every 3 weeks) for 3 cycles during the neoadjuvant treatment phase. Sintilimab will be administered as IV infusion 3 weeks during the post-operative adjuvant phase up to 1 year.
  Interventions: Drug: sintilimab

INTERVENTIONS:
Drug: IBI110 — R2PD d1 IV every 3 weeks
  Arms: IBI110+sintilimab
Drug: sintilimab — 200mg d1 IV every 3 weeks

SUMMARY:
The main purpose of this study is to evaluate the neoadjuvant therapy efficacy of IBI110 in combination with sintilimab versus sintilimab alone based on pathologic complete response (pCR) rate in stage IIB (primary tumor > 4 cm ) to IIIB (N2 only) subjects with radically resectable NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Have NSCLC that has been classified as stage IIB (primary tumor > 4 cm), IIIA, or IIIB (N2 only) per the 8th edition of TNM staging system of International Association for the Study of Lung Cancer (IASLC) and the American Joint Committee on Cancer (AJCC).
2. Subjects with non-squamous NSCLC should undergo genetic testing to confirm the absence of epidermal growth factor receptor (EGFR) sensitizing mutations or anaplastic lymphoma kinase (ALK) rearrangements;
3. Eligible for radical resection (R0 resection) at the thoracic surgeon's discretion, and the lung function meets the criteria for planned surgery;
4. Have at least one measurable lesion per RECIST v1.1 criteria;
5. Have a performance scale of 0 or 1 on the Eastern Cooperative Oncology Group Performance Status (ECOG PS)

Exclusion Criteria:

1. Have pathological evidence for small cell carcinoma, neuroendocrine carcinoma, sarcoma, lymphoepithelial rumen carcinoma, salivary gland tumor, or mesenchymal tumor from the biopsy.
2. Have been previously exposed to immune-mediated therapies, including but not limited to LAG-3 antibody drugs, anti-cytotoxic T lymphocyte antigen-4 (CTLA-4), anti-PD-1, anti-PD-L1, and anti-PD-L2 antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
pCR | Approximately 21 to 28 days after operation
  defined as having no residual visible tumor cells in the surgically resected primary tumor and lymph node samples (ypT0N0)
Incidence of serious adverse events (SAEs), treatment-emergent AEs (TEAEs) and immune-related AEs (irAEs) | up to 90 days after the last administration
  An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly/birth defect or is an important medical event that may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed before. A TEAE will be defined as any new AE that begins, or any pre-existing condition that worsens in severity, after at least 1 dose of study treatment has been administered. irAEs will be assessed.
Number of participants with abnormality in vital signs | up to 90 days after the last administration
  Blood pressure, pulse, respiratory rate, and temperature will be assessed.
Number of participants with abnormality in hematology parameters | up to 90 days after the last administration
  Blood samples will be collected to evaluate hemoglobin, mean corpuscular volume (MCV), white blood cell (WBC) count, platelets, 5-part differential white cell count, mean platelet volume and coagulation factors including international normalized ratio (INR), activated partial thromboplastin time (aPTT) and prothrombin time (PT).
Number of participants with abnormality in clinical chemistry parameters | up to 90 days after the last administration
  Blood samples will be collected to evaluate sodium, potassium, calcium, magnesium, chloride, glucose, creatinine, urea or blood urea nitrogen (BUN), bicarbonate, amylase, bilirubin, alkaline phosphatase, aspartate aminotransferase (AST), alanine aminotransferase (ALT), total protein, albumin, lactate dehydrogenase and lipase.
Number of participants with abnormality in clinical chemistry parameters | up to 90 days after the last administration
  Blood samples will be collected to evaluate sodium, potassium, calcium, magnesium, chloride, glucose, creatinine, urea or BUN, bicarbonate, amylase, bilirubin, alkaline phosphatase, AST, ALT, total protein, albumin, lactate dehydrogenase and lipase.
Number of participants with abnormality in routine urinalysis parameters | up to 90 days after the last administration
  Urine samples will be collected to evaluate specific gravity, leucocyte esterase, nitrite, blood, bilirubin, protein, glucose, ketones and urobilinogen.
Number of participants with abnormality in ECG parameters | up to 90 days after the last administration
  12-lead ECG will be obtained using an ECG machine. Participants will be in supine or a semi-recumbent position (about 30 degrees of elevation) and rested for approximately 2 minutes before ECGs are recorded.

SECONDARY OUTCOMES:
EFS （Event Free Survival） | up to 3 years
  defined as time from randomization to any of the following events: progression of disease that precludes surgery, local or distant recurrence, or death due to any cause
major pathological response (MPR) rate | Approximately 21 to 28 days after operation
  defined as ≤ 10% residual viable tumor cells in the surgically resected primary tumor and lymph nodes
radical resection (R0 resection) rate | Approximately 21 to 28 days after operation
  defined as free resection margins, systematic node dissection or sampling, and the highest mediastinal node negative for tumor
ORR （Objective Response rate,） | Within 7 days before surgery
  defined as the ratio of subjects who have achieved investigator assessed complete response (CR) and partial response (PR) per RECIST v1.1
OS （Overall Survival） | up to 3 years
  defined as the time from randomization to death from any cause
Immunogenicity | From date of randomization to 30 days after last dose of the drug
  includes the positive rate of anti-drug antibody (ADA) and neutralizing antibody (NAb) in subjects
maximum concentrations (Cmax ) | from first administration of IBI110 to 3 days before the operation
  Maximum serum concentration that IBI110 and Sintilimab achieves in the body after the drug has been administered and before the administration of a second dose.
the area under the drug plasma concentration-time curve (AUC) | from first administration of IBI110 to 3 days before the operation
  Area under the concentration-time curve from time zero to last measurable concentration (AUC)
half-life (t1/2) | from first administration of IBI110 to 3 days before the operation
  defined as the time it takes for the concentration of IBI110 and Sintilimab in the plasma or the total amount in the body to be reduced by 50%.
clearance (CL) | from first administration of IBI110 to 3 days before the operation
  a pharmacokinetic measurement of the volume of plasma from which IBI110 and Sintilimab are completely removed per unit time
volume of distribution (V). | from first administration of IBI110 to 3 days before the operation
  calculated by the amount of the drug in the body divided by the plasma concentration.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No